CLINICAL TRIAL: NCT06954714
Title: Late-lumen Changes After Drug-Coated Balloon Angioplasty Versus Drug-Eluting Stents in De Novo Coronary Lesions
Acronym: LARGER-DCB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Young Joon Hong, Professor, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNUH-2025-115
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease
Keywords: drug-coated balloon; intravascular ultrasound
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: prospective, multi-center, off-label, randomized controlled, non-inferiority trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug-eluting stent (Active Comparator): In DES group, latest second-generation DES will be used in accordance with standard practice guideline.
  Interventions: Procedure: Drug-eluting stent implantation
- Drug-coated balloon (Experimental): In DCB group, commercially available DCB (Agent, Boston Scientific, USA) will be used. DCB angioplasty will be recommended as follows to fully optimized procedural results. First, DCB size should be 1:1 ratio with reference vessel size. Second, delivery time of DCB should be within 30 seconds. Third, total inflation time of DCB will be recommended from 30 to 60 seconds.
  Interventions: Procedure: Drug-coated balloon angioplasty

INTERVENTIONS:
Procedure: Drug-eluting stent implantation — IVUS (OPTICROSS, Boston Scientific, USA) will be recommended to select proper size of predilatation balloon (semi- or non-compliant balloon), DCB, or DES. Optimal lesion preparation is defined as satisfying all of the followings: 1) a fully inflated balloon of the correct size for the vessel (balloon with vessel ratio >0.90); 2) ≤35% residual stenosis; 3) TIMI (Thrombolysis In Myocardial Infarction) flow grade 3; and 4) the absence of a flow-limiting coronary artery dissection.15 After successful lesion preparation, patients will receive either DCB or DES according to randomly allocated groups.
  In DES group, latest second-generation DES will be used in accordance with standard practice guideline.
  Arms: Drug-eluting stent
Procedure: Drug-coated balloon angioplasty — IVUS (OPTICROSS, Boston Scientific, USA) will be recommended to select proper size of predilatation balloon (semi- or non-compliant balloon), DCB, or DES. Optimal lesion preparation is defined as satisfying all of the followings: 1) a fully inflated balloon of the correct size for the vessel (balloon with vessel ratio >0.90); 2) ≤35% residual stenosis; 3) TIMI (Thrombolysis In Myocardial Infarction) flow grade 3; and 4) the absence of a flow-limiting coronary artery dissection.15 After successful lesion preparation, patients will receive either DCB or DES according to randomly allocated groups.
  In DCB group, commercially available DCB (Agent, Boston Scientific, USA) will be used. DCB angioplasty will be recommended as follows to fully optimized procedural results. First, DCB size should be 1:1 ratio with reference vessel size. Second, delivery time of DCB should be within 30 seconds. Third, total inflation time of DCB will be recommended from 30 to 60 seconds.
  Arms: Drug-coated balloon

SUMMARY:
This study aims to compare late-lumen loss (LLL) between DCB and DES to treat de novo coronary artery stenosis by intravascular ultrasound (IVUS).

DETAILED DESCRIPTION:
Drug-eluting stent (DES) is the standard of care for patients with coronary artery disease who are eligible for percutaneous coronary intervention (PCI).1 During long-term follow-up, remained metallic stent strut continuously related with stent-related cardiovascular events.2 As an alternative option to DES, drug-coated balloon (DCB) which has benefit of having shorter DAPT maintenance duration due to the absence of metallic scaffolds and polymers, has been introduced. Based on meta-analysis based on many randomized clinical trials (RCT),3,4 its use has been established in in-stent restenosis of bare-metal stents and DES.5 Furthermore, recent RCTs demonstrated efficacy and safety of DCB in de novo coronary lesions in small vessels with reference vessel size <3.0mm.6,7 For the patients with de novo, non-complex coronary artery lesions, REC-CAGEFREE I tested the non-inferiority of DCB angioplasty with DES implantation, irrespective of vessel diameter.8 Overall, 2272 patients were randomly assigned to the DCB or the DES group. At 2 years, adverse events occurred in 6.4% of DCB group and 3.4% of DES group and failed to prove the non-inferiority of DCB angioplasty (P for non-inferiority=0.65). Regarding the heterogenous results, it is questionable that DCB angioplasty for large de novo lesions is safe and effective compared with DES implantation.

On this background, the current study aims to compare late-lumen loss (LLL) between DCB and DES to treat de novo coronary artery stenosis by intravascular ultrasound (IVUS).

ELIGIBILITY:
Inclusion Criteria

1. Subject must be at least 19 years of age
2. Subject who is able to understand risks, benefits and treatment alternatives and sign informed consent voluntarily
3. Patients with at least one lesion with greater than 50% diameter stenosis or fractional flow reserve ≤0.80 requiring revascularization in de-novo coronary artery of reference vessel size ≥3.0 mm

Exclusion Criteria

1. Patients unable to provide consent
2. Patients with known intolerance to aspirin, P2Y12 inhibitors, or components of drug-eluting stents
3. Patients with angiographic findings of 1) Left main coronary artery disease 2) In-stent restenosis is the cause of target lesion 3) Target lesion in bypass graft 4) True bifurcation lesion that requires upfront 2-stenting
4. Patients who have non-cardiac co-morbid conditions with life expectancy <1 year
5. Patients who may result in protocol non-compliance (site investigator's medical judgment)
6. Patients with cardiogenic shock or cardiac arrest
7. Patients with severe left ventricular systolic dysfunction (ejection fraction <30%)
8. Patients with severe valvular heart disease requiring open heart surgery
9. Pregnant or lactating women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Late-lumen loss | 9 months after last patient enrollment
  Mean difference of late-lumen loss between DCB and DES in IVUS

SECONDARY OUTCOMES:
Minimal lumen diameter in QCA | 9 months after last patient enrollment
  Mean difference of minimal lumen diameter in QCA
% diameter stenosis in QCA | 9 months after last patient enrollment
  Mean difference of % diameter stenosis in QCA
Minimal lumen diameter in IVUS | 9 months after last patient enrollment
  Mean difference of minimal lumen diameter in IVUS
Cardiovascular death | 1 year after last patient enrollment
  Cardiovascular death
All-cause death | 1 year after last patient enrollment
  All-cause death
Rate of target vessel-MI | 1 year after last patient enrollment
  Target vessel-MI
Rate of non-fatal MI | 1 year after last patient enrollment
  Non-fatal MI
Rate of target lesion revascularization | 1 year after last patient enrollment
  Clinically indicated target lesion revascularization
Rate of target vessel revascularization | 1 year after last patient enrollment
  Clinically indicated target vessel revascularization
Rate of any revascularization | 1 year after last patient enrollment
  Any revascularization
Rate of vessel or stent thrombosis | 1 year after last patient enrollment
  Definite or probable thrombosis
Cardiovascular death or target vessel-related myocardial infarction | 1 year after last patient enrollment
  A composite of cardiovascular death or target vessel-related myocardial infarction
All-cause death or non-fatal MI | 1 year after last patient enrollment
  A composite of all-cause death or non-fatal myocardial infarction
Target vessel failure | 1 year after last patient enrollment
  A composite of cardiovascular death, target-vessel myocardial infarction, and clinically indicated target vessel revascularization
Target lesion failure | 1 year after last patient enrollment
  A composite of cardiovascular death, target-vessel myocardial infarction, and clinically indicated target lesion revascularization
Cardiovascular death, target-vessel MI, or vessel or stent thrombosis | 1 year after last patient enrollment
  A composite of cardiovascular death, target-vessel MI, or vessel or stent thrombosis
All-cause death, non-fatal myocardial infarction, or target vessel revascularization | 1 year after last patient enrollment
  A composite of all-cause death, non-fatal myocardial infarction, or target vessel revascularization
BARC type 2, 3, or 5 bleeding | 1 year after last patient enrollment
  BARC type 2, 3, or 5 bleeding
Cerebrovascular accident | 1 year after last patient enrollment
  Ischemic stroke, hemorrhagic stroke, or transient ischemic attack

CONTACTS AND LOCATIONS:
Overall Officials: Young Joon Hong, MD, PhD, Study Chair — Chonnam National University
Locations (9):
- South Korea (9):
  - Kosin University Gospel Hospital, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - Chonnam National University, Gwangju
  - Jeonbuk National University Hospital, Jeonju
  - Samsung Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Ulsan University Hospital, Ulsan
  - Yeosu Jeil Hospital, Yeosu

IPD SHARING:
Plan to Share IPD: Yes
Yes After publication of main paper, de-identified data will be shared upon reasonable requests after discussion by Executive Committee.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publication of main paper.
Access Criteria: Executive Committee will discuss to share the de-identified data upon reasonable requests.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-24): https://cdn.clinicaltrials.gov/large-docs/14/NCT06954714/Prot_SAP_000.pdf